CLINICAL TRIAL: NCT04139473
Title: Randomized Trial of Hepaticojejunostomy Versus Duct-to-duct Anastomosis in Right Lobe Living Donor Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Siu-Ho Chok, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 12-070
Record Dates: First submitted 2019-10-09; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepaticojejunostomy (Active Comparator): Patients undergo right lobe living donor liver transplantation will receive hepaticojejunostomy
  Interventions: Procedure: Hepaticojejunostomy / Duct-to-duct anastomosis
- Duct-to-duct anastomosis (Active Comparator): Patients undergo right lobe living donor liver transplantation will receive duct-to-duct anastomosis
  Interventions: Procedure: Hepaticojejunostomy / Duct-to-duct anastomosis

INTERVENTIONS:
Procedure: Hepaticojejunostomy / Duct-to-duct anastomosis

SUMMARY:
The scarcity of deceased donor organ supply has driven the practice of living donor liver transplantation (LDLT). Right lobe LDLT (RLDLT) has developed over the last 10 years to extend the benefit of LDLT to adult patients. With technical refinement, the results have significantly improved but bile duct complications remain the Achilles heel that affects the recipient's long-term outcome.Hepaticojejunostomy (HJ) was originally the standard technique for bile duct reconstruction in RLDLT but in recent years, duct-to-duct anastomosis (DDA) has been adopted by most transplant centers. The advantages of duct-to-duct reconstruction include a shorter operation time, less infection complications, more physiologic enteric functions and easier endoscopic access to the biliary tract but bile duct complication, particularly stricture is the major concern. The development of stricture is likely to be related to the blood supply of the anastomosis. We hypothesize that HJ has a better blood supply and is associated with a lower overall bile duct complication rate than duct-to-duct anastomosis. We propose a randomized trial to test this hypothesis and to compare various outcome measures between HJ and duct-to-duct reconstruction. The results of the study will set the standard for the technique of biliary reconstruction in RLDLT and will further advance this procedure.

DETAILED DESCRIPTION:
Liver transplantation is a life-saving procedure for patients with end-stage liver disease. The demand for the operation, however, always exceeds the supply from deceased organ donors and living donor liver transplant (LDLT) has been developed to provide an alternative option. LDLT was initially limited to paediatric recipients because of the restriction imposed by the graft size. In order to extend the benefit of LDLT to adult recipients, we proposed the use of a right lobe liver graft from a living donor and performed the first RLDLT for an adult recipient on May 9, 1996. Following the report of our first series of 8 cases in 1997, RLDLT has developed rapidly and has been adopted by many transplant programs around the world. LDLT has the most significant impact in Asia where the issue of organ shortage is most extreme. The availability of RLDLT for adult recipients provides the driving force for a drastic increase in LDLT in recent years. Our recent survey (unpublished data) indicated that the number of LDLT performed in Asia each year has increased by 9 folds since the introduction of RLDLT 10 years ago and is continuously rising. In the year 2005, LDLT accounts for 90% of the 1497 liver transplants performed in Asia (excluding mainland China). In Hong Kong, over two-thirds of the liver transplants are from living donors and the majority (90%) are RLDLT performed for adult recipients. RLDLT involved one of the most complicated and technically demanding surgical procedure. When our first series was reported in 1997, there was a high morbidity and reoperation rate in the recipients. Since then, various advances in technique and management have been introduced, including a better understanding of the minimum graft size requirement and anatomic variants of the right lobe, improved selection criteria for donors and recipients, as well as technical modifications; particularly in venous outflow and biliary reconstruction. There is a learning curve in RLDLT and through the lessons learnt in our first 100 RLDLT, we have dramatically improved the outcome of both the donors and recipients and an excellent graft survival rate of over 90% could be achieved even in high-risk recipients. The major technical hurdle that remains is biliary complication which affects the long-term outcome and quality of life and is occasionally the cause of graft loss and patient death. Hepaticojejunostomy was the standard technique for biliary reconstruction in RLDLT. The reported incidence of biliary complications in early reported retrospective series was high, ranging from 15 to 64%. Wach et al. first reported the technique of duct-to-duct reconstruction for RLDLT in 1998. Biliary stricture developed four weeks later and the anastomosis was subsequently revised to a Roux-e-Y HJ. Nonetheless, duct-to-duct reconstruction has the potential advantages of a shorter operation time, less septic complications, more physiologic enteric functions and easier endoscopic access to the biliary tract and these seem so obvious that duct-to-duct anastomsis has become the preferred technique in many transplant centers. In a retrospective study of 259 adult LDLTs; including 225 RLDLT from the Asan Medical Center in South Korea, Shin Hwang et al. reported an increasing preference for duct-to-duct anastomosis over HJ, with duct-to-duct anastomosis comprising 29.9% of the procedures in 2000 increasing to 69.3% in 2001 and 83.7% in 2002. The 3-year cumulative biliary complication rate, however, increased progressively form 13.7% in 2000 to 15.8% in 2001 and 25.4% in 2002. This rising incidence of biliary complication contrasted sharply with the improving results in other outcome measures of RLDLT which has been attributed to the learning curve effect. The authors demonstrated that for a right lobe graft with a single biliary reconstruction, a graft duct size less than 4 mm in diameter was a risk factor for biliary stricture in duct-to-duct anastomosis but not for HJ. They suggested that duct-to-duct anastomosis had inherent deficiencies that could not be overcome by current surgical techniques and recommended HJ as the preferred approach under such circumstances.We performed a retrospective study at our centre, in 265 RLDLT recipients, 55 (20.8%) developed postoperative BAS. The BAS rates were 21.4% (43/201) for recipients undergoing duct-to-duct anastomosis during transplantation, 18.9% (10/53) for recipients undergoing HJ, and 18.2% (2/11) for recipients undergoing both procedures. BAS and non-BAS patients had comparable demographics. The number of graft bile duct openings (P = 0.516) and the size of the graft's smallest bile duct (5 versus 5 mm, P = 0.4) were not significantly different between BAS and non-BAS patients. Univariate analysis showed that the factors associated with postoperative BAS were the recipient warm ischemia time (55 versus 51 minutes, P = 0.026), graft cold ischemia time (120 versus 108 minutes, P = 0.046), stent use (21.8% versus 7.1%, P = 0.001), postoperative acute cellular rejection (29.1% versus 11.0%, P = 0.001), and University of Wisconsin solution use (21.8% versus 7.1%, P = 0.001). Multivariate analysis showed that the cold ischemia time (odds ratio = 1.012, 95% confidence interval = 1.002-1.023, P = 0.014) and acute rejection (odds ratio = 3.180, 95% confidence interval = 1.606-6.853, P = 0.002) were significant factors. The graft survival rates of BAS and non-BAS patients were comparable. One patient required retransplantation for secondary biliary cirrhosis. In conclusion, BAS remains common after adult RLDLT regardless of DDA or HJ. The graft cold ischemia time and postoperative acute cellular rejection are significantly associated with postoperative BAS. A randomised controlled trial is definitely needed to see which methoid is superior to another. Since we reported the first series of RLDLT in 1997, we have introduced numerous technical refinements; particularly in venous outflow and biliary reconstruction. HJ was originally the standard technique and technical modifications were directed at preserving the blood supply to the graft right hepatic duct during the donor operation. A retrospective study on the first 74 right lobe transplants showed that the biliary complication rate has decreased significantly from 43% in the first 37 patients to 8% only in the second 37 patients. In particular, there was no biliary leakge in the second group of patients. Since then, however, we have switched from HJ to duct-to-duct anastomosis as the preferred technique for biliary reconstruction because of its apparently obvious advantages. With the new technique, however, three of 41 patients (7%) had biliary leakage and 10 (24%) developed biliary stricture at a median of 5.8 months (range 1.5 to 16.9 months) after transplant. These results were comparable to those of the Kyoto group in which the incidence of bile leakage was 10% and that of stricture 23%. A randomized trial is the only way to objectively determine whether HJ or duct-to-duct anastomosis should be the preferred technique for biliary reconstruction in RLDLT. Since the results of biliary reconstruction is highly dependent on the technique of the surgical team, a multi-center study would introduce a serious surgeons' variable that may compromise the interpretation of the results. Hence a randomized trial in a single high volume center using a standard technique by a single surgical team would be the best approach.

ELIGIBILITY:
Inclusion Criteria:

* recipient age older than 18 years
* primary transplant

Exclusion Criteria:

* recipient refusal/withdrawal
* haemodynamic instability at the time of biliary reconstruction
* biliary reconstruction with duct-to-duct anastomosis is unsafe or technically not feasible
* unhealthy recipient's bile duct, anatomical variant in donor's right duct
* biliary reconstruction with hepaticojejunostomy is unsafe or technically not feasible
* excessively edematous bowel, failure to create Roux-en-Y jejunal loop due to excessive
* bowel adhesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-05-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Biliary complications | 5 years
  Compare all biliary-associated complications after operation including leakage and stricture

SECONDARY OUTCOMES:
Operative time for liver transplantation | intraoperative
  Duration of operative time
Gastrointestinal function after liver transplantation | 5 years
  Return of gastrointestinal function
Hospital stay after liver transplantation | 5 years
  Duration of hospital stay
Chances of re-intervention | 5 years
  Re-intervention rate

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo CM, Fan ST, Liu CL, Lo RJ, Lau GK, Wei WI, Li JH, Ng IO, Wong J. Extending the limit on the size of adult recipient in living donor liver transplantation using extended right lobe graft. Transplantation. 1997 May 27;63(10):1524-8. doi: 10.1097/00007890-199705270-00027. PMID 9175822
- [Background] Lo CM, Fan ST, Liu CL, Wei WI, Lo RJ, Lai CL, Chan JK, Ng IO, Fung A, Wong J. Adult-to-adult living donor liver transplantation using extended right lobe grafts. Ann Surg. 1997 Sep;226(3):261-9; discussion 269-70. doi: 10.1097/00000658-199709000-00005. PMID 9339932
- [Background] Wachs ME, Bak TE, Karrer FM, Everson GT, Shrestha R, Trouillot TE, Mandell MS, Steinberg TG, Kam I. Adult living donor liver transplantation using a right hepatic lobe. Transplantation. 1998 Nov 27;66(10):1313-6. doi: 10.1097/00007890-199811270-00008. PMID 9846514
- [Background] Marcos A, Fisher RA, Ham JM, Shiffman ML, Sanyal AJ, Luketic VA, Sterling RK, Posner MP. Right lobe living donor liver transplantation. Transplantation. 1999 Sep 27;68(6):798-803. doi: 10.1097/00007890-199909270-00012. PMID 10515380
- [Background] Trotter JF, Wachs M, Everson GT, Kam I. Adult-to-adult transplantation of the right hepatic lobe from a living donor. N Engl J Med. 2002 Apr 4;346(14):1074-82. doi: 10.1056/NEJMra011629. No abstract available. PMID 11932476
- [Background] Malago M, Testa G, Frilling A, Nadalin S, Valentin-Gamazo C, Paul A, Lang H, Treichel U, Cicinnati V, Gerken G, Broelsch CE. Right living donor liver transplantation: an option for adult patients: single institution experience with 74 patients. Ann Surg. 2003 Dec;238(6):853-62; discussion 862-3. doi: 10.1097/01.sla.0000098619.71694.74. PMID 14631222
- [Background] Todo S, Furukawa H, Jin MB, Shimamura T. Living donor liver transplantation in adults: outcome in Japan. Liver Transpl. 2000 Nov;6(6 Suppl 2):S66-72. doi: 10.1053/jlts.2000.19009. PMID 11084089
- [Background] Bak T, Wachs M, Trotter J, Everson G, Trouillot T, Kugelmas M, Steinberg T, Kam I. Adult-to-adult living donor liver transplantation using right-lobe grafts: results and lessons learned from a single-center experience. Liver Transpl. 2001 Aug;7(8):680-6. doi: 10.1053/jlts.2001.26509. PMID 11510011
- [Background] Lee SG, Park KM, Hwang S, Lee YJ, Kim KH, Ahn CS, Choi DL, Joo SH, Jeon JY, Chu CW, Moon DB, Min PC, Koh KS, Han SH, Park SH, Choi GT, Hwang KS, Lee EJ, Chung YH, Lee YS, Lee HJ, Kim MH, Lee SK, Suh DJ, Kim JJ, Sung KB. Adult-to-adult living donor liver transplantation at the Asan Medical Center, Korea. Asian J Surg. 2002 Oct;25(4):277-84. doi: 10.1016/S1015-9584(09)60192-5. PMID 12470999
- [Background] Nakamura T, Tanaka K, Kiuchi T, Kasahara M, Oike F, Ueda M, Kaihara S, Egawa H, Ozden I, Kobayashi N, Uemoto S. Anatomical variations and surgical strategies in right lobe living donor liver transplantation: lessons from 120 cases. Transplantation. 2002 Jun 27;73(12):1896-903. doi: 10.1097/00007890-200206270-00008. PMID 12131684
- [Background] Olthoff KM, Merion RM, Ghobrial RM, Abecassis MM, Fair JH, Fisher RA, Freise CE, Kam I, Pruett TL, Everhart JE, Hulbert-Shearon TE, Gillespie BW, Emond JC; A2ALL Study Group. Outcomes of 385 adult-to-adult living donor liver transplant recipients: a report from the A2ALL Consortium. Ann Surg. 2005 Sep;242(3):314-23, discussion 323-5. doi: 10.1097/01.sla.0000179646.37145.ef. PMID 16135918
- [Background] Lo CM, Fan ST, Liu CL, Chan JK, Lam BK, Lau GK, Wei WI, Wong J. Minimum graft size for successful living donor liver transplantation. Transplantation. 1999 Oct 27;68(8):1112-6. doi: 10.1097/00007890-199910270-00009. PMID 10551638
- [Background] Fan ST, Lo CM, Liu CL. Technical refinement in adult-to-adult living donor liver transplantation using right lobe graft. Ann Surg. 2000 Jan;231(1):126-31. doi: 10.1097/00000658-200001000-00018. PMID 10636112
- [Background] Lo CM, Fan ST, Liu CL, Wong J. Hepatic venoplasty in living-donor liver transplantation using right lobe graft with middle hepatic vein. Transplantation. 2003 Feb 15;75(3):358-60. doi: 10.1097/01.TP.0000046527.19422.3E. PMID 12589159
- [Background] Fan ST, Lo CM, Liu CL, Tso WK, Wong J. Biliary reconstruction and complications of right lobe live donor liver transplantation. Ann Surg. 2002 Nov;236(5):676-83. doi: 10.1097/00000658-200211000-00019. PMID 12409675
- [Background] Lo CM, Fan ST, Liu CL, Yong BH, Wong Y, Lau GK, Lai CL, Ng IO, Wong J. Lessons learned from one hundred right lobe living donor liver transplants. Ann Surg. 2004 Jul;240(1):151-8. doi: 10.1097/01.sla.0000129340.05238.a0. PMID 15213631
- [Background] Liu CL, Lo CM, Chan SC, Fan ST. Safety of duct-to-duct biliary reconstruction in right-lobe live-donor liver transplantation without biliary drainage. Transplantation. 2004 Mar 15;77(5):726-32. doi: 10.1097/01.tp.0000116604.89083.2f. PMID 15021836
- [Background] Hwang S, Lee SG, Sung KB, Park KM, Kim KH, Ahn CS, Lee YJ, Lee SK, Hwang GS, Moon DB, Ha TY, Kim DS, Jung JP, Song GW. Long-term incidence, risk factors, and management of biliary complications after adult living donor liver transplantation. Liver Transpl. 2006 May;12(5):831-8. doi: 10.1002/lt.20693. PMID 16528711
- [Background] Yi NJ, Suh KS, Cho JY, Kwon CH, Lee KU. In adult-to-adult living donor liver transplantation hepaticojejunostomy shows a better long-term outcome than duct-to-duct anastomosis. Transpl Int. 2005 Nov;18(11):1240-7. doi: 10.1111/j.1432-2277.2005.00209.x. PMID 16221154
- [Background] Ishiko T, Egawa H, Kasahara M, Nakamura T, Oike F, Kaihara S, Kiuchi T, Uemoto S, Inomata Y, Tanaka K. Duct-to-duct biliary reconstruction in living donor liver transplantation utilizing right lobe graft. Ann Surg. 2002 Aug;236(2):235-40. doi: 10.1097/00000658-200208000-00012. PMID 12170029
- [Background] Grewal HP, Shokouh-Amiri MH, Vera S, Stratta R, Bagous W, Gaber AO. Surgical technique for right lobe adult living donor liver transplantation without venovenous bypass or portocaval shunting and with duct-to-duct biliary reconstruction. Ann Surg. 2001 Apr;233(4):502-8. doi: 10.1097/00000658-200104000-00004. PMID 11303131